CLINICAL TRIAL: NCT05804357
Title: The Effect of Manual Therapy on Psychological Factors and Quality of Life in Lumbal Disc Herniation Patients: A Single Blind Randomized Clinical Study
Brief Title: The Effect of Manual Therapy on Psychological Factors and Quality of Life in Lumbal Disc Herniation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10879717-016.18.22
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Intervertebral Disc Displacement; Lumbar Disc Herniation; Psychological; Quality of Life
Keywords: Lumbar disc herniation; Manual therapy; Kinesiophobia; Anxiety and depression; Pain catastrophe
MeSH Terms: conditions — Intervertebral Disc Displacement; Kinesiophobia; Anxiety Disorders; Depression | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Intervention Model Description: This study was designed as a double-blind randomized controlled clinical trial. In order to carry out the prospectively designed study, ethics committee approval was obtained from the Non-Interventional Clinical Research Ethics Committee of Muş Alparslan University with the decision numbered 21 taken at the meeting dated 29.12.2020 and numbered 15. Informed consent was obtained from all patients included in the study before the study.
Who Masked: Participant
Masking Description: Eligible patients were divided into two groups using the closed envelope method at a ratio of 1:1. The patients did not know which group they were in. Mobilization applications and other clinical tests were performed by the same physiotherapist in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): In our study, stabilization exercises were applied to the patients in the exercise group. The treatment was applied two days a week for five weeks, for a total of ten sessions. After the end of the treatment, stabilization exercises were recommended as a home exercise program until the follow-up evaluation at the third month. A telephone connection was established with the patients once a week and the home program was followed up.Stabilization exercises: It is an approach that is combined with diaphragmatic breathing and activates the passive. The stabilization exercise program was applied in three phases and was progressed in line with the developments in the patients
  Interventions: Behavioral: Exercise
- Manual Therapy Group (Experimental): In our study, stabilization exercises and spinal mobilization practices were performed to the patients in the manual therapy group. The treatment was applied two days a week for five weeks, for a total of ten sessions. After the end of the treatment, stabilization exercises were recommended as a home exercise program until the follow-up evaluation at the third month. A telephone connection was established with the patients once a week and the home program was followed up.Mobilization applications were applied at Maitland IV degree as standard.Three mobilization methods were applied Anterior-Posterior Lumbal Spinal Mobilization Lumbal Spinal Rotational Mobilization Joint Mobilization in Lumbal Flexion Position
  Interventions: Behavioral: Manual Therapy

INTERVENTIONS:
Behavioral: Manual Therapy — Mobilization applications are passive movements that do not involve pushing or stimuli, applied within the range of motion or up to the physiological range of motion
  Other Names: Lumbal Spinal Mobilization
  Arms: Manual Therapy Group
Behavioral: Exercise — It is an approach that is combined with diaphragmatic breathing, activating the passive-active musculoskeletal and neural systems. In this approach, transversus abdominis and multifudus muscles are activated as deep core muscles.
  Other Names: Stabilization Exercise
  Arms: Exercise Group

SUMMARY:
When the literature is examined, there are studies examining the relationship between low back pain and anxiety depression, quality of life and LDH in patients with lumbar disc herniation. There are many studies on the clinical use of manual therapy methods in LDH. Most of these studies examine the effect of manual therapy on pain and functional level. However, there are hardly any studies examining the effect of manual therapy on quality of life and psychological factors in LDH patients.

The aim of our study is to examine the effect of mobilization, which is a manual therapy application, on psychological factors (kinesiophobia, pain catastrophic thought, anxiety and depression) and quality of life in LDH patients.

DETAILED DESCRIPTION:
There are various treatment options that can be applied to patients with lumbar disc herniation (LDH). These are basically divided into 2 categories: surgical and conservative treatment. Conservative treatment methods in the treatment of LDH aim to prevent the disease from transitioning to interventional methods and / or surgical treatment and to improve the complaints that negatively affect the quality of life. Conservative treatment; It includes informing the patient, bed rest, drug treatments, exercise, thermotherapy, electrotherapy, traction, orthoses, back school and manual therapy applications. Manual therapy; It is used to reduce pain, provide joint and tissue mobility, inhibit sympathetic reflex activity, normalize muscle tone and dissolve adhesions. Manual therapy is the manual treatment of the spine with two different applications such as manipulation and mobilization.

The clinical effects of manual therapy in LDH patients were examined. The aim of this study was to investigate the effect of manual therapy on psychological factors and quality of life in patients with lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* It was determined as being diagnosed with LDH by MR by a physical therapy physician
* Having pain of at least 3 levels or more according to the Visual Analogue Scale
* Being between the ages of 18-65.

Exclusion Criteria:

* History of spinal surgery
* History of autoimmune disease (ankylosing spondylitis, rheumatoid arthritis or other)
* Spondylolysis and spondylolisthesis
* Spinal fracture
* Heart pathology
* History of stroke,
* Cauda equina syndrome
* Continuous use of pain medication
* Spinal inflammation,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | The change of pain assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  McGill-Melzack Pain Questionnaire :It is a questionnaire applied to determine the location, characteristics, relationship with time and severity of low back pain. The total score is obtained by summing the points corresponding to the answer given according to each category. While the maximum score was 78, the minimum score was set to 0. The higher the pain, the higher the score.

SECONDARY OUTCOMES:
Anxiety and Depression Assessment | The change of anxiety and depression assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Hospital Anxiety and Depression Scale :It is a self-assessment scale applied to determine the risk of anxiety and depression in the patient, to measure its level and change in severity. It contains a total of 14 questions, seven of which measure anxiety and the other seven measure depression.
Kinesiophobia Assessment | The change of anxiety and depression assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Tampa Kinesiophobia Scale :Consisting of 17 questions, the scale measures individuals' fear of re-injury with movement. The questions in the scale are calculated with the Likert scoring type consisting of 4 points. Patients are given a minimum score of 17 and a maximum score of 68. The high score obtained as a result of the scale indicates the high degree of kinesiophobia. In studies, 37 points and above are defined as high kinesiophobia.
Pain Catastrophizing Assessment | The change of pain catastrophe assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Pain Catastrophizing Scale: It reliably assesses certain variables, such as fears, feelings or thoughts, severe pain, disability, and emotional disturbances associated with individuals' past pain experiences. The scale consists of 13 questions scored between 0-4 (0=Never, 1=A little. 2=Moderately, 3=Seriously, 4=Always). An increase in the scale score indicates a high fear of experiencing pain.
Quality of Life Assessment | The change of quality of life assessed before treatment, through treatment completion, an average of 1 week and during follow-up 3 months after treatment
  Nottingham Health Profile (NHP): It is a valid-reliable quality of life scale used to evaluate the physical, emotional and social effects of diseases on individuals. It consists of six sections, including pain, physical activity, energy, sleep, social isolation and emotional reaction, and a total of 38 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Taşkaya, Principal Investigator — Muş Alparslan University
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taskaya B, Taskent I, Cakilli M, Yilmaz O. The Effect of Manual Therapy on Psychological Factors and Quality of Life in Lumbar Disc Herniation Patients: A Single Blinded Randomized Clinical Trial. Int J Environ Res Public Health. 2024 Sep 18;21(9):1234. doi: 10.3390/ijerph21091234. PMID 39338117